CLINICAL TRIAL: NCT04034810
Title: Safety and Efficacy of Silk Vista and Silk Vista Baby Flow Diverter for Intracranial Aneurysm Treatment, an Observational, Prospective, Single Arm, International, Multicenter Study.
Brief Title: Safety and Efficacy of Silk Vista and Silk Vista Baby Flow Diverter for Intracranial Aneurysm Treatment
Acronym: FIRST
Status: Active, not recruiting | Type: Observational
Sponsor: Balt Extrusion (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP 201802 SILK VISTA
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Intracranial Aneurysm; Flow Diverter
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intracranial aneurysm treated with Silk vista and silk vista baby — Patients with intracranial aneurysm(s) intended to be treated with the silk vista and silk vista baby according to standard of care.

SUMMARY:
The FIRST study is an observational, prospective, multi-center, international, single-arm, study. The aim of the study is to collect safety and efficacy information on the use of the silk vista and silk vista baby flow diverter in order to assess clinical safety and performance of the device for treating intracranial aneurysms.

All patients with intracranial aneurysm ruptured or unruptured, whatever the localization of the aneurysm, and treated with silk vista or silk vista baby, will be consecutively enrolled in the study.

The patient's inclusion and follow up in the study will occur as part of their usual standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with intracranial aneurysms intended to be treated with the silk vista and silk vista baby (decision of use silk vista and silk vista baby is done independently and prior to the participation of the patient in the study)
2. Patients with recanalized aneurysms previously treated with coils exclusively are also eligible.
3. In case of multiple aneurysms, only treatment with silk vista and silk vista baby are allowed (between the initial index procedure to the 12 months follow up visit)
4. Patient ≥ 18 years, who signed an informed consent.

Exclusion Criteria:

1. Patient presenting with contra-indications to the use of silk vista and silk vista babyaccording to the IFU (Instruction for Use).
2. Recanalized aneurysms initially treated with stent (including stent assisted coiling)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an intracranial aneurysm treated with silk vista and silk vista baby.
Sampling Method: Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Morbi-mortality of silk vista and silk vista baby in the treatment of intracranial aneurysms. | At 12-months (-3 / + 6 months) post procedure
  Characterized by the rate of the permanent neurologic deficits and procedure related mortality.
Morbi-mortality of silk vista and silk vista baby in the treatment of intracranial aneurysms. | At 12-months (-3 / + 6 months) post procedure
  Characterized by the clinical outcome assessed by mRS of the permanent neurologic deficits and procedure related mortality.

SECONDARY OUTCOMES:
Safety of silk vista and silk vista baby | At T0
  Assessed by the rate of adverse events
Safety of silk vista and silk vista baby | At hospital discharge
  Assessed by the rate of adverse events
Safety of silk vista and silk vista baby | Up to 30 days (-10 / + 21 days) post- procedure.
  Assessed by the rate of adverse events
Safety of silk vista and silk vista baby | At 6 months (-2/+3 months) post- procedure.
  Assessed by the rate of adverse events
Safety of silk vista and silk vista baby | At 12 months (-3/+6 months) post- procedure.
  Assessed by the rate of adverse events
Safety of silk vista and silk vista baby | At 3 years post procedure
  Assessed by the rate of adverse events
Safety of silk vista and silk vista baby | At 5 years post procedure
  Assessed by the rate of adverse events
Efficacy of silk vista and silk vista baby | At T0
  Assessed by aneurysm occlusion rate
Efficacy of silk vista and silk vista baby | At hospital discharge
  Assessed by aneurysm occlusion rate
Efficacy of silk vista and silk vista baby | Up to 30 days (-10 / + 21 days) post- procedure.
  Assessed by aneurysm occlusion rate
Efficacy of silk vista and silk vista baby | Up to 6 months (-2/+3 months) post- procedure
  Assessed by aneurysm occlusion rate
Efficacy of silk vista and silk vista baby | Up to 12 months (-3 / + 6 months) post procedure
  Assessed by aneurysm occlusion rate
Efficacy of silk vista and silk vista baby | Up to 3 years post procedure
  Assessed by aneurysm occlusion rate
Efficacy of silk vista and silk vista baby | Up to 5 years post procedure
  Assessed by aneurysm occlusion rate
Technical procedure | At T0
  The practices related to the use of silk vista baby will be describe

CONTACTS AND LOCATIONS:
Overall Officials: Mario Martinez Galdamez, Dr, Principal Investigator — Hospital Clinico Universitario de Valladolid (HCUV), Spain
Locations (29):
- Universitätsklinik für Neurologie, Salzburg, Austria
- CHC Saint Joseph Liège, Liège, Belgium
- University Hospital Centre Zagreb, Zagreb, Croatia
- France (13):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Hopital Cavale Blanche, Brest
  - Hospices Civils de Lyon - Hôpital Neurologique, Bron
  - CHU Caen, Radiologie interventionelle, Caen
  - Centre Hospitalier Universitaire Clermont Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Grenoble Alpes, Grenoble
  - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Chu Dupuytren Limoges, Limoges
  - Hôpital Privé Clairval, Marseille
  - Fondation Rothschild, Paris
  - Pitié-Salpêtrière Hospital, Paris
  - CHU Chalre Nicolle, Rouen
  - Centre Hospitalier Régional Universitaire de Tours, Tours
- Munich LMU University, München, Germany
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
- Italy (4):
  - Niguarda Hospital, Milan
  - San Gerardo Hospital, Monza
  - Cà Foncello Hospital, Treviso
  - Santa maria della misericordia hospital, Udine
- Radboud University medical Center, Nijmegen, Netherlands
- Spain (5):
  - Hospital Universitario de cruces, Barakaldo
  - Ramon y Cajal hospital, Madrid
  - Hopsital universidad puerta de hierro, Madrid
  - Unversitario Central de Asturias, Oviedo
  - Hospital Clinico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No